CLINICAL TRIAL: NCT06852534
Title: Probing the Role of Feature Dimension Maps in Visual Cognition: Expt 1.1 (Behavioral)
Brief Title: Probing the Role of Feature Dimension Maps in Visual Cognition: Impact of Salience Level (Eye-tracking Follow-up Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Santa Barbara (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5-24-0700: Expt 1.1 Behavioral; R01EY035300 (NIH)
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Basic Science: Visual Attention in Healthy Participants; Attention

STUDY DESIGN:
Masking Description: Participants will typically be unaware of the conditions presented, though because these involve manipulations of stimuli or task demands, they may be aware of the manipulation. This is not expected to impact the primary outcome measures (e.g., behavioral performance).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manipulations of graded feature salience (Expt 1.1) (Experimental): Participants will view stimuli made salient based on feature contrast in one feature dimensions (color or motion direction; or checkerboard luminance contrast). The degree to which a location is salient will be manipulated based on the feature contrast across multiple values
  Interventions: Other: Stimulus properties: salience-defining feature; Other: Stimulus properties: magnitude of salience

INTERVENTIONS:
Other: Stimulus properties: salience-defining feature — The feature used to define a salient location will be varied across trials (checkerboard contrast; motion direction; color hue)
Other: Stimulus properties: magnitude of salience — The magnitude of the salient location will be varied across trials independently from salience-defining feature (based on feature contrast)

SUMMARY:
How does one know what to look at in a scene? Imagine a "Where's Waldo" game - it's challenging to find Waldo because there are many 'salient' locations in the picture, each vying for one's attention. One can only attend to a small location on the picture at a given moment, so to find Waldo, one needs to direct their attention to different locations. One prominent theory about how one accomplishes this claims that important locations are identified based on distinct feature types (for example, motion or color), with locations most unique compared to the background most likely to be attended. An important component of this theory is that individual feature dimensions (again, color or motion) are computed within their own 'feature maps', which are thought to be implemented in specific brain regions. However, whether and how specific brain regions contribute to these feature maps remains unknown.

The goal of this study is to determine how brain regions that respond strongly to different feature types (color and motion) and which encode spatial locations of visual stimuli extract 'feature dimension maps' based on stimulus properties, including feature contrast. The investigators hypothesize that feature-selective brain regions act as neural feature dimension maps, and thus encode representations of salient location(s) based on their preferred feature dimension. The investigators will collect eye-tracking data while participants view visual stimuli made salient based on different combinations of feature dimensions. From the eye-tracking data, the investigators will construct fixation heat maps on the feature dimensions for all levels of salience, allowing them to connect behavioral data to the latter fMRI dataset. Each participant will freely view the stimuli as they appear on the computer display. Across trials, the investigators will manipulate 1) the 'strength' of the salient locations based on how different the salient stimulus is compared to the background, 2) the number of salient locations, and 3) the feature value(s) used to make each location salient. Altogether, these manipulations will help the investigators fully understand these critical salience computations in the healthy human visual system.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 55 years of age
* normal or corrected-to-normal vision

Exclusion Criteria:

* N/A

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Gaze position | Through study completion, an average of one week
  The investigators will use the measured gaze position in (x,y) coordinates to reconstruct fixations to stimuli on various levels of salience throughout the trials.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Sprague, Principal Investigator — University of California, Santa Barbara
Locations (1):
- University of California, Santa Barbara, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw eye-tracking data will be shared with researchers immediately upon publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available indefinitely beginning with publication of results
Access Criteria: Raw behavioral/eyetracking data will be publicly available on the lab's Open Science Framework page (https://osf.io/ufjzl/), and analysis code will be available on GitHub (an online tool for storing and managing code; github.com/SpragueLab)
URL: https://osf.io/ufjzl/

REFERENCES:
- [Background] Mackey WE, Winawer J, Curtis CE. Visual field map clusters in human frontoparietal cortex. Elife. 2017 Jun 19;6:e22974. doi: 10.7554/eLife.22974. PMID 28628004
- [Background] Hallenbeck GE, Sprague TC, Rahmati M, Sreenivasan KK, Curtis CE. Working memory representations in visual cortex mediate distraction effects. Nat Commun. 2021 Aug 5;12(1):4714. doi: 10.1038/s41467-021-24973-1. PMID 34354071
- [Background] Sprague TC, Itthipuripat S, Vo VA, Serences JT. Dissociable signatures of visual salience and behavioral relevance across attentional priority maps in human cortex. J Neurophysiol. 2018 Jun 1;119(6):2153-2165. doi: 10.1152/jn.00059.2018. Epub 2018 Feb 28. PMID 29488841
- [Background] Sprague TC, Adam KCS, Foster JJ, Rahmati M, Sutterer DW, Vo VA. Inverted Encoding Models Assay Population-Level Stimulus Representations, Not Single-Unit Neural Tuning. eNeuro. 2018 Jun 5;5(3):ENEURO.0098-18.2018. doi: 10.1523/ENEURO.0098-18.2018. eCollection 2018 May-Jun. No abstract available. PMID 29876523
- [Background] Sprague TC, Boynton GM, Serences JT. The Importance of Considering Model Choices When Interpreting Results in Computational Neuroimaging. eNeuro. 2019 Dec 20;6(6):ENEURO.0196-19.2019. doi: 10.1523/ENEURO.0196-19.2019. Print 2019 Nov/Dec. PMID 31772033
- [Background] Laumann TO, Gordon EM, Adeyemo B, Snyder AZ, Joo SJ, Chen MY, Gilmore AW, McDermott KB, Nelson SM, Dosenbach NU, Schlaggar BL, Mumford JA, Poldrack RA, Petersen SE. Functional System and Areal Organization of a Highly Sampled Individual Human Brain. Neuron. 2015 Aug 5;87(3):657-70. doi: 10.1016/j.neuron.2015.06.037. Epub 2015 Jul 23. PMID 26212711
- [Background] Allen EJ, St-Yves G, Wu Y, Breedlove JL, Prince JS, Dowdle LT, Nau M, Caron B, Pestilli F, Charest I, Hutchinson JB, Naselaris T, Kay K. A massive 7T fMRI dataset to bridge cognitive neuroscience and artificial intelligence. Nat Neurosci. 2022 Jan;25(1):116-126. doi: 10.1038/s41593-021-00962-x. Epub 2021 Dec 16. PMID 34916659
- [Background] Fedorenko E. The early origins and the growing popularity of the individualsubject analytic approach in human neuroscience. Current Opinion in Behavioral Sciences. 2021; 40:105-112.
- [Background] Naselaris T, Allen E, Kay K. Extensive sampling for complete models of individual brains. Current Opinion in Behavioral Sciences. 2021; 40:45-51.
- [Background] Poldrack RA. Diving into the deep end: a personal reflection on the MyConnectome study. Current Opinion in Behavioral Sciences. 2021; 40:1-4.
- [Background] Pritschet L, Taylor CM, Santander T, Jacobs EG. Applying dense-sampling methods to reveal dynamic endocrine modulation of the nervous system. Curr Opin Behav Sci. 2021 Aug;40:72-78. doi: 10.1016/j.cobeha.2021.01.012. Epub 2021 Feb 25. PMID 35369044
- [Background] Gratton C, Nelson SM, Gordon EM. Brain-behavior correlations: Two paths toward reliability. Neuron. 2022 May 4;110(9):1446-1449. doi: 10.1016/j.neuron.2022.04.018. PMID 35512638
- [Background] Smith PL, Little DR. Small is beautiful: In defense of the small-N design. Psychon Bull Rev. 2018 Dec;25(6):2083-2101. doi: 10.3758/s13423-018-1451-8. PMID 29557067
- [Background] Sprague TC, Serences JT. Attention modulates spatial priority maps in the human occipital, parietal and frontal cortices. Nat Neurosci. 2013 Dec;16(12):1879-87. doi: 10.1038/nn.3574. Epub 2013 Nov 10. PMID 24212672
- [Background] Itthipuripat S, Vo VA, Sprague TC, Serences JT. Value-driven attentional capture enhances distractor representations in early visual cortex. PLoS Biol. 2019 Aug 9;17(8):e3000186. doi: 10.1371/journal.pbio.3000186. eCollection 2019 Aug. PMID 31398186
- [Background] Poltoratski S, Tong F. Resolving the Spatial Profile of Figure Enhancement in Human V1 through Population Receptive Field Modeling. J Neurosci. 2020 Apr 15;40(16):3292-3303. doi: 10.1523/JNEUROSCI.2377-19.2020. Epub 2020 Mar 5. PMID 32139585
- [Background] Poltoratski S, Ling S, McCormack D, Tong F. Characterizing the effects of feature salience and top-down attention in the early visual system. J Neurophysiol. 2017 Jul 1;118(1):564-573. doi: 10.1152/jn.00924.2016. Epub 2017 Apr 5. PMID 28381491